CLINICAL TRIAL: NCT02266940
Title: A Phase 1, Open Label, Randomised, Single Dose, Three Way Crossover Study to Explore the Relative Bioavailability of DS 1971a Given as a 200 mg Tablet Formulation and a 200 mg Oral Suspension, and to Explore the Effects of Administration With a High Fat Meal on the Relative Bioavailability of the Tablet Formulation
Brief Title: Relative Bioavailability DS-1971a Suspension and Tablets and Food Effect on DS-1971a Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DS1971-A-E104
Record Dates: First submitted 2014-10-09; First posted 2014-10-17 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2015-01

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — DS-1971a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 200mg DS-1971a oral suspension fasted (Experimental): 200 mg DS 1971a given as oral suspension in fasted condition
  Interventions: Drug: DS-1971a suspension
- 200 mg DS-1971a tablet fasted (Experimental): single 200 mg DS 1971a oral tablet in fasted condition
  Interventions: Drug: DS-1971a tablet
- 200 mg DS-1971a tablet fed (Experimental): single 200 mg DS 1971a oral tablet given in fed condition
  Interventions: Drug: DS-1971a tablet

INTERVENTIONS:
Drug: DS-1971a suspension — DS 1971a will be supplied as a powder or crystals and prepared at the study site for administration as an oral suspension with a taste masking agent.
  Arms: 200mg DS-1971a oral suspension fasted
Drug: DS-1971a tablet — A 200 mg DS 1971a tablet for oral administration
  Arms: 200 mg DS-1971a tablet fasted; 200 mg DS-1971a tablet fed

SUMMARY:
This is an open label, randomised, 3 treatment, 3 period crossover study. This study is designed to assess the relative bioavailability of DS 1971a from a tablet formulation and a reconstituted oral suspension and the effect of a high fat meal on the relative bioavailability of DS 1971a from the tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 65 years, inclusive
* Subjects must be in good general health as determined by medical history, physical examination and screening investigations, and be taking no regular medication
* A body mass index (BMI) in the range 18 to 30 kg/m^2, inclusive, and weighing between 50 and 100 kg. BMI is calculated as weight [kg]/(height [m])^2
* Female subjects must be of nonchildbearing potential as follows:

Must be postmenopausal (the last menstrual period was at least 12 months before Screening, and a follicle stimulating hormone [FSH] test at Screening confirms postmenopausal status); or Must be surgically sterile having undergone hysterectomy, bilateral oophorectomy, bilateral salpingectomy and/or bilateral tubal ligation

* Willing and able to consume a standard Food and Drug Administration (FDA) high fat meal
* Willing to comply with all study restrictions, including the use of contraception, concomitant medication, and dietary and lifestyle restrictions
* Sufficient intelligence to understand the nature of the study and any hazards of participating in it. Ability to communicate satisfactorily with the Investigator and to participate in, and comply with the requirements of, the entire study
* Have given written consent to participate after reading the information and consent form, and after having the opportunity to discuss the study with the Investigator or his/her delegate
* Have given written consent to have his/her data entered into The Over-volunteering Prevention System (TOPS)

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, ECG findings, or laboratory values that could interfere with the objectives of the study or the safety of the subject
* Presence of or history of acute or chronic illness, including (but not limited to) liver or kidney disease, hypertension, seizures, or any known impairment of endocrine, or other specific body-organ dysfunction
* Presence or history of severe adverse reaction to any medicine
* Presence or history of malignant disease
* Acute or chronic infectious disease, including human immunodeficiency virus (HIV), hepatitis B virus (HBV) or C virus (HCV) infection
* Surgery (eg, stomach bypass) or medical condition that might affect absorption of medicines
* Significant illness within 4 weeks before the dose of study medication
* Participation in another clinical study of a new chemical entity or a prescription medicine within the previous 3 months, or unwilling to abstain from participating in other clinical studies during the study and for 3 months after receipt of their final dose of study medication
* Participation in another clinical study with DS-1971a
* Blood pressure (BP) and heart rate in semi supine position at the screening examination outside the ranges 90-140 mmHg systolic, 40-90 mmHg diastolic; heart rate 40-100 beats/min. Subjects with Stage 1 hypertension (systolic 140 160 mmHg; diastolic 90 100 mmHg) may be enrolled provided they do not have evidence of end organ damage, diabetes or a 10 year cardiovascular risk >20%
* Estimated glomerular filtration rate (eGFR) <80 mL/min/1.73m^2 or an absolute creatinine value above the upper limit of normal (ULN). eGFR will be estimated at Screening using the modification of diet in renal disease (MDRD) equation
* Abnormal ECG waveform morphology at Screening that would preclude accurate measurement of the QT interval duration
* Corrected QT interval (Fridericia's formula) (QTcF) interval duration >430 msec for men or >450 msec for women, obtained as an average from the measurements on duplicate screening ECGs
* Use of any prescription medicine or over-the-counter (OTC) medications, herbal remedies (such as St John's Wort), or food known to be strong inhibitors or strong inducers of cytochrome (CYP) enzymes (also known as CYP450 enzymes) during the 30 days before the dose of study medication; use of any other prescription or OTC medicine, including dietary supplements or herbal remedies, during the 7 days before the first dose of study medication
* Consumption of certain foods or beverages before the dose and throughout the study period
* Loss of more than 400 mL blood during the 3 months before the study, eg, as a blood donor
* Abuse of drugs or alcohol during the 2 years before the first dose of study medication, or intake of more than 21 units of alcohol weekly (for men) or 14 units of alcohol weekly (for women)
* Use of tobacco products or nicotine containing products during the 3 months before the dose of trial medication
* Likely possibility that the volunteer will not cooperate with the requirements of the protocol
* Objection by General Practitioner (GP) to volunteer entering the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics profile of DS-1971a | 3 days from dose administration
  Plasma concentration time data will be analysed using non compartmental methods. The following PK parameters will be estimated: Cmax, Tmax and AUClast. If data permit, AUC0-inf, CL/F, Vd/F and T½ will be estimated.

SECONDARY OUTCOMES:
number and severity of adverse events as a measure of safety and tolerability | administration of first dose to 10 weeks
  number and severity of adverse events as a measure of safety and tolerability
changes in clinical laboratory profile | administration of first dose to 10 weeks
  haematology, biochemistry, and urinalysis
changes in physical exam profile | administration of first dose to 10 weeks
  Physical examination profile includes; Height and weight, heart rate, blood pressure (BP), oral temperature and respiration rate, 12 lead electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/